CLINICAL TRIAL: NCT03419065
Title: Relaxation Interventions for Pre-term Mothers on Hospitalized Bed-Rest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Towson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 09-A052R3
Record Dates: First submitted 2017-12-01; First posted 2018-02-01 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: High Risk Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Relaxation Intervention (Other): Women hospitalized on bed-rest for high risk pregnancy participated in Relaxation Interventions.
  Interventions: Behavioral: Relaxation Intervention

INTERVENTIONS:
Behavioral: Relaxation Intervention — Relaxing Music combined with Progressive Muscle relaxation and guided imagery

SUMMARY:
The purpose of this study is to investigate the effects of participation in relaxation exercises on pregnant women who are hospitalized on bed-rest.

DETAILED DESCRIPTION:
Women, 18 or older, who consent to this study will participate in a preliminary interview. Study participants will then be trained in the use of progressive muscle relaxation and guided imagery for pregnancy. Participants will be issued a listening device and an audio file and asked to practice it on a daily basis while in the hospital.

Prior to discharge or delivery, the participant will be visited by a member of the research team who will conduct a follow-up interview. The interviews and the relaxation practice sessions will take between 30 and 45 minutes each. The interviews will be audio-recorded, although no identifying information about the participants will be recorded.

At the conclusion of the study, participants will be given a CD of the audio relaxation program and thanked for their participation in the study.

There is minimal risk anticipated in association with participation in this study. All information gained from this study will remain confidential and is for educational purposes only. Participants are entitled to terminate their participation in the study at any time.

It is hoped that the results of this study will provide information about an intervention that may be beneficial to women with high-risk pregnancies. It is also hoped that participation in the exercises will be enjoyable and/or beneficial to you in some way. The results of this study may be used to justify further studies or to influence the type of interventions offered in this or similar settings.

All data collected from the research will remain confidential. Data collected from participants will immediately be assigned an identification number so that no one will be able to identify any individuals in the study.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women on bed rest for high risk pregnancy

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2013-06-01 (Actual); Study Completion 2013-06-01 (Actual)

PRIMARY OUTCOMES:
Interview | 5-7 days
  Participants participated in a follow up interview

SECONDARY OUTCOMES:
Post-survey | 5-7 days
  Participants completed a brief post-survey

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Yeager, PhD, OTR/L, Principal Investigator — Towson University
Locations (1):
- Towson University, Towson, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
de-identified data may be shared through publication but no identifying information will be shared